CLINICAL TRIAL: NCT02372032
Title: Percutaneous Lumbar Discectomy (PLD) Combined With Ozone Versus Percutaneous Lumbar Discectomy (PLD) for Treatment of Lumbar Disc Herniation:A Single-Blind Prospective Randomized Controlled Trial
Brief Title: A Trial of Percutaneous Lumbar Discectomy Combined With Ozone for Treatment of LDH
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Gao-jun Teng, Professor of Radiology & Chair,Department of Radiology, Zhongda Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014ZDSYLL134
Record Dates: First submitted 2015-02-06; First posted 2015-02-26 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Lumbar Disc Herniation
Keywords: Herniation; Discectomy; Ozone
MeSH Terms: conditions — Intervertebral Disc Displacement; Hernia

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- PLD combined with ozone (Experimental): Patients diagnosed as lumbar disc herniation undergoing percutaneous lumbar discectomy combined with ozone therapy.
  Interventions: Procedure: percutaneous lumbar discectomy; Procedure: ozone therapy
- pure PLD (Active Comparator): Patients diagnosed as lumbar disc herniation undergoing percutaneous lumbar discectomy(PLD).
  Interventions: Procedure: percutaneous lumbar discectomy

INTERVENTIONS:
Procedure: percutaneous lumbar discectomy — process percutaneous lumbar discectomy
Procedure: ozone therapy — percutaneous intradiscal ozone injection
  Arms: PLD combined with ozone

SUMMARY:
Lumbar disc herniation (LDH) is a common pathological process leading to spinal surgery. Open discectomy used to be a widespread procedure for surgical treatment for symptomatic LDH. Currently, several minimal invasive surgeries have been uesd widely. Percutaneous lumbar discectomy(PLD) and ozone therapy are two widely used minimal invasive treatment, and ozone therapy combined other minimally invasive treatment could improve other minimally invasive treatment's clinical effectiveness. The effectiveness of which has been proved to be comparable to conventional open discectomy.

In this study, a single-blind randomized controlled trial will be performed to evaluate the effectiveness of two minimal invasive discectomy, percutaneous lumbar discectomy combined with ozone and percutaneous lumbar discectomy, for the treatment of symptomatic LDH.

Two groups of patients will be investigated; 1) patients diagnosed with lumbar disc herniation undergoing PLD combined with ozone, and 2) patients diagnosed with lumbar disc herniation undergoing PLD.

The primary endpoints of the study will be changes in in pain and functional status by the Visual Analog Scale (VAS) and functional status as measured by Oswestry Low Back Disability Questionnaire (Oswestry Disability Index,ODI) and Japanese Orthopaedic Association (JOA) as measured at pre- and post-operation, 1 month, 3 months, 6 months. Secondary outcomes include response evaluation by MacNab response evaluation criteria as measured at pre- and post-operation, 1 month, 3 months, 6 months. Treatment effect is defined as the difference in the mean change from baseline between the two groups.

For the first time,the results of this trial will provide scientific evidence as to the relative effectiveness of PLD combined with ozone versus PLD for minimal invasive surgical treatment for symptomatic lumbar disc herniation.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 years.
* 4 or more weeks low back pain and/or lower-limb radiation pain.
* MRI and/or CT test confirm diagnosis lumbar disc herniation and level(s).
* Invalid after Non-steroidal anti-inflammatory medical therapy and physical therapy.
* Pain level（Visual Analog Scale）≥5.

Exclusion Criteria:

* Spinal tumors.
* Spine infections, fractures, slippage(more than I °) and other deformities.
* Combining with spinal stenosis, lateral recess stenosis, yellow ligament hypertrophy.
* Nucleus pulposus herniated too much, dural sac compressed more than 50%;
* Psychological, cognitive disorders which may affect the reliability of the outcome;
* Previous lumbar disc surgery;
* Bleeding tendency or severe cardiovascular disease can not tolerate surgery;
* Don't accept the trial's informed consent;
* Possible pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in Visual Analog Scale(VAS) | Baseline, post-op 1 month, 3 months, 6 months
Changes from baseline in Oswestry Low Back Disability Questionnaire(ODI) | Baseline, post-op 1 month, 3 months, 6 months
Changes from baseline in Japanese Orthopaedic Association Scores(JOA) | Baseline, post-op 1 month, 3 months, 6 months

SECONDARY OUTCOMES:
Response evaluation measured by MacNab criteria | post-op 1 month, 3 months, 6 months
  Response evaluation as measured by MacNab criteria

CONTACTS AND LOCATIONS:
Overall Officials: Gao-jun Teng, Ph.D,MD, Principal Investigator — Zhongda Hospital
Locations (1):
- Zhongda Hospital,Southeast University, Nanjing, Jiangsu, China